CLINICAL TRIAL: NCT06334198
Title: The Effect of Naldemedine on Opioid-induced Bowel Dysfunction. An Investigator Initiated, Randomized, Double-blinded, Placebo-controlled, Cross-over Clinical Trial
Brief Title: The Effect of Naldemedine on Opioid-induced Bowel Dysfunction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asbjørn Mohr Drewes (Other)
Responsible Party: Sponsor-Investigator, Asbjørn Mohr Drewes, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Naldemedine_OIBD; 2023-507744-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Opioid-Induced Bowel Dysfunction; Constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — naldemedine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): Naldemedine + tramadol
  Interventions: Drug: Naldemedine; Drug: Tramadol
- Placebo treatment (Placebo Comparator): Placebo + tramadol
  Interventions: Drug: Placebo; Drug: Tramadol

INTERVENTIONS:
Drug: Naldemedine — Naldemedine is administered orally once daily in the morning in a dosage of 0.2 mg.
  Arms: Active treatment
Drug: Placebo — Placebo is administered orally once daily in the morning.
  Arms: Placebo treatment
Drug: Tramadol — In both arms, tramadol is administered orally twice daily in a dosage of 100 mg (daily total of 200mg).

SUMMARY:
Opioid-induced bowel dysfunction is a frequent condition during opioid therapy for chronic pain. Indeed, up to 90% of people on opioid treated patients experience constipation. Standard laxative treatment is often ineffective in opioid-induced constipation, but peripheral acting mu-receptor antagonists (PAMORAs) have the potential to block the effects of opioids in the gastrointestinal tract while preserving the central analgesic effect. In this study, we will investigated the effects of Naldemedine in preventing the development of opioid-induced bowel dysfunction and constipation during treatment with tramadol

ELIGIBILITY:
Inclusion Criteria:

* Healthy (assessed by a study-affiliated medical doctor)
* Signed informed consent
* Able to read and understand Danish.
* Male (to avoid influence of menstrual cycles).
* Northern European descent (to minimize genetic variance influences on drug metabolism).
* The researcher believes that the participant understands the study details, is compliant and is expected to complete the study.
* Opioid naïve (no history of opioid use/addiction. Opioid use more than a year ago to treat pain post-surgery is accepted. Opioid use in connection with participation in a clinical trial more than a year ago is accepted)
* Between 20 and 40 years of age.
* A STAI (Spielberger State-Trait Anxiety Inventory) score in the range of 20-37 i.e., classified as "no or low anxiety" at inclusion.

Exclusion Criteria:

Known hypersensitivity or allergy towards the used pharmaceutical compounds or pharmaceutical compounds similar to those used in the study.

* Less than three spontaneous bowel movements per week.
* Participation in other studies within 14 days prior to first visit.
* Expected need of medical/surgical treatment during the study.
* Any diagnosed disease, which investigator concludes will affect the trial (including all contraindicated complications: severe chronic obstructive pulmonary disease, pulmonary heart disease, severe bronchial asthma, paralytic ileus, hypercapnia, serious respiratory depression with hypoxia, moderate to severe decreased liver function, gastrointestinal obstruction or perforation, acute surgical abdominal complications such as appendicitis, Mb. Crohn's, ulcerative colitis, and toxic mega colon).

History of substance abuse (alcohol, tetrahydrocannabinol, benzodiazepine, central stimulants and/or opioids, urine drug test will be performed prior to treatment start).

* History of major mental disorders (e.g., major anxiety, major depression or treatment with psychoactive medications etc.)
* Metal implants or pacemaker.
* Daily use of prescription only medicine
* Daily alcohol consumption
* Participation motivated by "wrongful" reasons such as poor economy or psychosocial issues e.g., problems in the family, loneliness, sadness. People with such problems may be more likely to develop substance dependence*.
* Intake of alcohol within 48 hours before start of study period or any alcohol consumption during each study period. If consumption takes place during the study the participant will be excluded.
* Use of any analgesic medication within 48 hours before start as well as for the duration of the study. If consumption takes place during the study the participant will be excluded.
* Nicotine use

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Total gastrointestinal transit time | From day 4 to day 8
  Difference in hours from ingestion of a 3D Transit Capsule to expulsion of the capsule during active and placebo treatment
Colorectal transit time | From day 4 to day 8
  Difference in hours from the entering in the colon of a 3D Transit Capsule to expulsion of the capsule during active and placebo treatment

SECONDARY OUTCOMES:
Constipation symptoms | From day 1 to day 10
  Measured on the Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire (ranging from 0 (symptom absent) to 4 (very severe).
Bowel movement frequency | From day 1 to day 10
  Number of spontaneous bowel movements per day
Stool consistency | From day 1 to day 10
  Rated on the Bristol Stool Form Scale (ranging from type 1 (constipation) - type 7 (diarrhea))
Gastrointestinal symptoms | Day 1 and day 10
  Measured on the Gastrointestinal Symptom Rating Score (GSRS) questionnaire (ranging from 0 (no discomfort) to 6 (very severe discomfort)
Opioid-induced constipation | Day 1 and day 10
  Measured by the Bowel Function Index (BFI) questionnaire (ranging from 0 (not at all) to 100 (very strong).
Diagnostic evaluation of opioid-induced constipation | Day 10
  Assessed using the Rome IV C6 criteria
Colonic motility patterns | From day 4 to day 8
  Number of motility patterns in the colon measured by the 3D Transit Capsule
Opiate withdrawal symptoms | Day 13, 14 or 15
  Measured by the Subjective Opiate Withdrawal Scale (ranging from 0 (not at all) to 4 /extremely)
Colon volume | Day 10
  Volumetric quantification of the colon measured using T2-weighted MRI images
Colonic water content | Day 10
  Analysis of colonic water content measured using heavily T2-weighted MRI images
Defecation assessment | Day 1 and day 10
  Analysis of rear-front pressure during a simulated defecation using the Fecobionics device

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Mohr Drewes, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark